CLINICAL TRIAL: NCT00602849
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalency Study of Sertraline Tablets 100 mg Under Fasting Conditions
Brief Title: Bioequivalency Study of Sertraline Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SERT-01
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sertraline

SUMMARY:
The objective of this study was the bioequivalence of a Roxane Laboratories' Sertraline Tablets, 100 mg, to Zoloft® Tablets, 100 mg (Pfizer) under fasting conditions using a single-dose, 2-treatment, 2-period, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* Treatment with any triptan within 30 days prior to or during the study.
* History of allergic or adverse response to sertraline or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2003-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Fourteen day washout

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Fly, Quebec, Canada